CLINICAL TRIAL: NCT01423318
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Study of the Safety, Tolerability, and Pharmacokinetics of Subcutaneous Doses of Lebrikizumab in Healthy Japanese and Caucasian Volunteers
Brief Title: A Study of Lebrikizumab in Healthy Japanese and Caucasian Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GB25741
Record Dates: First submitted 2011-08-22; First posted 2011-08-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — lebrikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Experimental)
  Interventions: Drug: lebrikizumab
- B (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: lebrikizumab — Dose-level cohorts receiving single subcutaneous dose
  Arms: A
Drug: placebo — single dose subcutaneously
  Arms: B

SUMMARY:
This randomized, double-blind, placebo-controlled, parallel-group study will evaluate the safety and pharmacokinetics of subcutaneous lebrikizumab in healthy Japanese volunteers. Healthy Japanese and Caucasian volunteers will be randomized to receive a single subcutaneous dose of either lebrikizumab or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy males and females, 18 to 55 years of age inclusive
* Caucasian, Japanese, or non-Japanese subjects. Caucasian or non-Japanese subjects will have no parents or grandparents of Japanese descent; Japanese subjects must be first, second or third generation
* Body weight between 45 and 105 kg, inclusive
* In good health, determined by no clinically significant findings from medical history, 12-lead ECG, vital signs, and laboratory evaluations
* Fertile males and women of childbearing potential must use appropriate form of contraception from screening until 60 days after study completion
* Negative for hepatitis B, hepatitis C, and HIV infection
* Negative for selected drugs of abuse at screening (not including alcohol) and at check-in (including alcohol)

Exclusion Criteria:

* Pregnant and lactating women
* History of clinically significant drug allergy and/or a known hypersensitivity to the study drug or formulation components
* History of helminthic infection or travel within the past 3 months to areas of high risk for parasitic exposure
* Use of prescription drugs including inhaled, oral, or parenteral corticosteroids and/or beta agonists, within 7 days prior to dosing or during the study
* Use of tobacco- or nicotine-containing products from 7 days prior to check-in, resulting in urinary cotinine >500 ng/mL. Minimal/intermittent smoking will be permitted during the study
* Participation in any other investigational drug trial in which receipt of an investigational study drug occurred within 30 days or 5 half-lives, whichever is longer, prior to check-in (Day -1)
* History of significant, chronic, or recurrent infections requiring treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events in healthy Japanese subjects | 120 days
Pharmacokinetics in healthy Japanese subjects: Area under the concentration-time curve (AUC) | 120 days

SECONDARY OUTCOMES:
Comparison of safety (incidence of adverse events) in healthy Japanese and Caucasian subjects | approximately 5 months
Comparison of pharmacokinetics (AUC) in healthy Japanese and Caucasian subjects | approximately 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (1):
- Honolulu, Hawaii, United States